CLINICAL TRIAL: NCT05713513
Title: Pilot Study to Manufacture Clinical T-cell Products for Future Treatment
Brief Title: Manufacture of Clinical T-cell Products for Future Treatment
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: PB_2018-00081; am23Khanna2
Record Dates: First submitted 2023-01-16; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Virus-specific T Cells
Keywords: T cell immunity; adoptive T cell therapy; Good Manufacturing Practice (GMP); leukapheresis
MeSH Terms: interventions — Leukapheresis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Leukapheresis — Leukapheresis to isolate 1x10e9 cells, examined for purity and specificity under Good Manufacturing Practice (GMP)

SUMMARY:
The aim of this pilot study is to validate the manufacture of T-cell products using GMP-approved reagents for future clinical use. Lymphocytes from whole blood of max 300ml from volunteers or from total 9 volunteer apheresates will be isolated to validate the protocol under Good Manufacturing Practice (GMP).

DETAILED DESCRIPTION:
Viral diseases occur in up to 50% of patients after transplantation. In most cases, there is a reactivation of the virus, which can be found latent or dormant in the body's own cells. The main reason for the occurrence of these diseases is the limited T-cell immunity, which serves to control these viruses in healthy people. To date, there are few effective and, depending on the virus, no established therapies. In addition, the established therapies are often associated with considerable toxicity. An alternative therapy, which has already shown success in the 1990s, is the administration of virus-specific T cells. Adoptive T cell therapies for the major pathogens emerging post-transplant are intended to use. In order to be used as therapy these cells must be manufactured under Good Manufacturing Practice (GMP). Leukapheresis from whole blood of maximum 300ml is used to generate the virus-specific T cells. These cells are examined for purity and specificity and are used for scientific purposes only. The aim of this study is to validate the manufacture of T-cell products using GMP-approved reagents for future clinical use.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* Immunoglobulins (Ig) G available for Epstein-Barr virus (EBV) or cytomegalovirus (CMV)
* Detectable T-cell response for EBV or CMV measured by flow cytometry (> 0.01%)

Exclusion Criteria:

* Infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) or human T-cell lymphoma virus (HTLV)-I/II

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The probands are selected on a voluntary basis. They are not directly involved in the project and take part in the study voluntarily. They either come from other working groups in the Department of Biomedicine or from the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Leukapheresis for manufacturing of T cell products by Good Manufacturing Practice (GMP) | one time assessment during the procedure
  Number of leukapheresis to isolate 1x10e9 cells for manufacturing of T cell products by Good Manufacturing Practice (GMP)
Purity after isolation defined as > 40% interferon-gamma positive cells | one time assessment during the procedure
  Purity after isolation defined as > 40% interferon-gamma positive cells

CONTACTS AND LOCATIONS:
Overall Officials: Nina Khanna, Prof. Dr. med., Principal Investigator — University Hospital Basel, Departement Infektiologie & Spitalhygiene
Locations (1):
- University Hospital Basel, Departement Infektiologie & Spitalhygiene, Basel, Switzerland